CLINICAL TRIAL: NCT05494983
Title: Pain, Sleep and Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PAIN,SLEEP,MICROBIOTA
Record Dates: First submitted 2022-06-22; First posted 2022-08-10 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sensitization, Central; Peripheral Sensitization; Gut Microbiota; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Session 1 : Peripheral Session (left) - session 2 Central Session (right) (Other): The susceptibility to develop peripheral sensitization will be assessed at the first experimental session, the stimulation will occur at the left forearm.
  The susceptibility to develop central sensitization will be assessed at the second experimental session, the stimulation will occur at the right forearm.
  In both experimental sessions, participants will have to fill questionnaires about the use of medications, the Stanford Sleepiness Scale, the Leeds Sleep Evaluation Questionnaire, and the first part of the State and Trait Anxiety Questionnaire. During sensory stimulation, an infrared camera will be used to measure pupil diameter which constitute an indirect correlate of stimulus-evoked phasic variations in activity of the locus coeruleus. In order to measure autonomic reactivity to pain stimuli, the heart rate variability will be measured by recording electrocardiography.
  Interventions: Other: Screening visit; Other: Peripheral sensitization session; Other: Central sensitization session
- Session 1 : Peripheral Session (right) - session 2 Central Session (left) (Other): The susceptibility to develop peripheral sensitization will be assessed at the first experimental session, the stimulation will occur at the right forearm.
  The susceptibility to develop central sensitization will be assessed at the second experimental session, the stimulation will occur at the left forearm.
  In both experimental sessions, participants will have to fill questionnaires about the use of medications, the Stanford Sleepiness Scale, the Leeds Sleep Evaluation Questionnaire, and the first part of the State and Trait Anxiety Questionnaire. During sensory stimulation, an infrared camera will be used to measure pupil diameter which constitute an indirect correlate of stimulus-evoked phasic variations in activity of the locus coeruleus. In order to measure autonomic reactivity to pain stimuli, the heart rate variability will be measured by recording electrocardiography.
  Interventions: Other: Screening visit; Other: Peripheral sensitization session; Other: Central sensitization session
- Session 1 : Central Session (left) - session 2 Peripheral Session (right) (Other): The susceptibility to develop central sensitization will be assessed at the first experimental session, the stimulation will occur at the left forearm.
  The susceptibility to develop peripheral sensitization will be assessed at the second experimental session, the stimulation will occur at the right forearm.
  In both experimental sessions, participants will have to fill questionnaires about the use of medications, the Stanford Sleepiness Scale, the Leeds Sleep Evaluation Questionnaire, and the first part of the State and Trait Anxiety Questionnaire. During sensory stimulation, an infrared camera will be used to measure pupil diameter which constitute an indirect correlate of stimulus-evoked phasic variations in activity of the locus coeruleus. In order to measure autonomic reactivity to pain stimuli, the heart rate variability will be measured by recording electrocardiography.
  Interventions: Other: Screening visit; Other: Peripheral sensitization session; Other: Central sensitization session
- Session 1 : Central Session (right) - session 2 Peripheral Session (left) (Other): The susceptibility to develop central sensitization will be assessed at the first experimental session, the stimulation will occur at the right forearm.
  The susceptibility to develop peripheral sensitization will be assessed at the second experimental session, the stimulation will occur at the left forearm.
  In both experimental sessions, participants will have to fill questionnaires about the use of medications, the Stanford Sleepiness Scale, the Leeds Sleep Evaluation Questionnaire, and the first part of the State and Trait Anxiety Questionnaire. During sensory stimulation, an infrared camera will be used to measure pupil diameter which constitute an indirect correlate of stimulus-evoked phasic variations in activity of the locus coeruleus. In order to measure autonomic reactivity to pain stimuli, the heart rate variability will be measured by recording electrocardiography.
  Interventions: Other: Screening visit; Other: Peripheral sensitization session; Other: Central sensitization session

INTERVENTIONS:
Other: Screening visit — The participants will be screened for inclusion and exclusion criteria and will be asked to fill the following questionnaires : Pittsburgh Sleep Quality Index, State and Trait Anxiety Questionnaire, Pain Catastrophizing Scale Fear of Pain Questionnaire, Perceived Stress Scale, Beck Depression Inventory, and questionnaires to assess their health status and the use of medications. A blood sample (to measure pro- and anti-inflammatory cytokines and perform metabolomic analyses) will be obtained. Enrolled participants will be given a wearable actimeter to assess daily total sleep duration during one week before the first experimental session. They will also be requested to complete daily a sleep diary during one week before each experimental session, and a food diary before the first experimental session. A fecal sample (to assess gut microbiota composition and perform metabolomic analyses) will be collected between the screening visit and the first experimental session.
Other: Peripheral sensitization session — The extent of neurogenic inflammation induced by topical capsaicin will be used as a measure of the susceptibility to sensitize at peripheral level. A solution of capsaicin will be applied to the skin of the left or right volar forearm for 30 minutes. The capsaicin-induced neurogenic inflammation can be quantified by assessing the intensity, extent and duration of the capsaicin-induced cutaneous flare response using thermal infrared imaging. Using heat stimuli delivered to the treated skin and surrounding skin, the intensity and duration of the capsaicin-induced hyperalgesia will also be assessed. The experimental session will last approximately two hours.
Other: Central sensitization session — The extent of secondary mechanical hyperalgesia induced by high-frequency electrical stimulation (HFS) of the skin of the left or right volar forearm will be used as a measure of the susceptibility to develop central sensitization. The stimulation will be delivered using a multi-pin electrode designed to preferentially activate epidermal free nerve endings. The strength, spatial extent and duration of the HFS-induced changes in pinprick sensitivity will be characterized by using calibrated mechanical pinprick stimuli. The experimental session will last approximately one hour.

SUMMARY:
The objective of this study in healthy volunteers is to evaluate whether the composition of the gut microbiota and sleep quality influence the susceptibility to develop peripheral and central sensitization of pain pathways.

In two different experimental sessions, the following factors will be tested: the influence of the composition of the gut microbiota on the susceptibility to develop peripheral sensitization of nociceptors, and the susceptibility to develop central sensitization of pain pathways. To assess susceptibility to peripheral sensitization, a solution of capsaicin (the active component of chili pepper) will be applied to the skin to induce neurogenic inflammation produced by the release of substances from nociceptors at the peripheral level. This neurogenic inflammation is characterized by a transient redness of the skin that will be measured with an infrared camera. To evaluate the susceptibility to sensitization at the central level, a high frequency electrical stimulation will be applied to the skin. This stimulation induces an increase in sensitivity to mechanical stimulation secondary to central sensitization. The intensity, extent and duration of this mechanical hyperalgesia will therefore be used as a measure of susceptibility to central sensitization.

A stool sample and a blood sample will be taken. These samples will be used to characterize the composition of the intestinal microbiota, as well as the metabolites produced by this microbiota. These analyses will allow a comparison of the composition of the microbiota and the metabolites in subjects with a tendency to develop low vs. high sensitization at the peripheral and central levels.

Similarly, sleep quality and average sleep duration will be assessed using questionnaires and a measurement of the participant's activity using a wrist movement sensitive bracelet. This information will be used to assess whether some of the interindividual variability in developing peripheral or central sensitization might be related to differences in sleep quality.

Finally, systemic inflammation could be a factor modulated by sleep and gut microbiota, influencing pain perception and susceptibility to sensitization. For this reason, systemic pro- and anti-inflammatory cytokines will be measured in the blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Ability to provide written informed consent
* Understanding French

Exclusion Criteria:

* Current or recent (< 2 months) use of antibiotics, probiotics, fiber supplements or any other molecule that modifies intestinal transit.
* Current or recent (< 1 month) use of non-steroidal anti-inflammatory drugs and glucocorticoids
* Not willing or able to abstain from acute alcohol intoxication from 7 days prior to each of the two study sessions.
* Consumption of alcohol 24 hours prior to each of the two study sessions.
* Consumption of hypnotics, centrally-acting analgesics or psychotropic drugs.
* Obesity: body mass index > 30 kg.m-2
* Pregnancy and breast-feeding
* Diabetes
* Cancer
* History of inflammatory bowel disease
* History of weight-loss surgery (e.g., gastric bypass, gastric band)
* History of autoimmune disease (e.g., lupus, rheumatoid arthritis)
* Evidence for any other clinically significant disease on direct questioning.
* Being a volleyball player due to risk of modified sensitivity of the volar forearm skin.
* Any implanted medical device such as cardiac pacemakers, cochlear implants and medication pumps.
* Dermatological condition affecting the skin of the volar forearms.
* History of an allergy to chili peppers/capsaicin.
* Any other reason to exclude the subject according to judgment by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between composition of the intestinal microbiota and its metabolites and the susceptibility of sensitization at the peripheral and central levels. | one week
  A stool sample and a blood sample will be taken. These samples will be used to characterize the composition of the intestinal microbiota, as well as the metabolites produced by this microbiota. These analyses will allow a comparison of the composition of the microbiota and the metabolites in subjects with a tendency to develop low vs. high sensitization at the peripheral and central levels.
  The gut microbiota composition will be analyzed using 16S rDNA sequencing. Untargeted metabolite profiling, in fecal and blood samples, will be performed using liquid chromatography (LC) coupled with tandem mass spectrometry (MS-MS) platforms.
Correlation between sleep quality and the susceptibility of sensitization at the peripheral and central levels. | five weeks
  Sleep quality will be assessed using questionnaires and a measurement of the participant's sleep using a wrist movement sensitive bracelet. This information will be used to assess whether some of the inter-individual variability in developing peripheral or central sensitization might be related to differences in sleep quality.
Correlation between sleep duration and the susceptibility of sensitization at the peripheral and central levels. | five weeks
  Average sleep duration will be assessed using questionnaires and a measurement of the participant's sleep using a wrist movement sensitive bracelet. This information will be used to assess whether some of the inter-individual variability in developing peripheral or central sensitization might be related to differences in sleep duration.

SECONDARY OUTCOMES:
Correlation between levels of systemic pro- and anti-inflammatory cytokines measured by multiplex assays and the susceptibility of sensitization at the peripheral and central levels. | one week
  Systemic inflammation could be an important factor modulated by sleep and the gut microbiota, influencing nociception and sensitization at peripheral and central levels. Plasma concentrations (pg/mL) of several pro-inflammatory (TNFa, IL-6, IL-1b, MCP-1) and anti-inflammatory (IL-10) markers will me measured using commercially available multiplex assays.
Correlation between pupil diameter and the susceptibility of sensitization at the peripheral and central levels. | five weeks
  During sensory stimulation, an infrared camera will be used to measure pupil diameter which has been shown to constitute an indirect correlate of stimulus-evoked phasic variations in activity of the locus coeruleus.
Correlation between heart rate variability and the susceptibility of sensitization at the peripheral and central levels. | five weeks
  In order to measure autonomic reactivity to pain stimuli, the heart rate variability will be measured by recording electrocardiography during experimental sessions.

CONTACTS AND LOCATIONS:
Overall Officials: André Mouraux, MD, PhD, Principal Investigator — UCLouvain, IONS
Locations (1):
- UCLouvain, IONS, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No